CLINICAL TRIAL: NCT05255991
Title: A Randomized, Double-blind, Placebo-controlled, Multinational, Phase 3 Study of the Efficacy and Safety of Inhaled Treprostinil in Subjects With Idiopathic Pulmonary Fibrosis (TETON-2)
Brief Title: Multinational Study of Efficacy and Safety of Inhaled Treprostinil in Subjects With Idiopathic Pulmonary Fibrosis
Acronym: TETON-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIN-PF-303; 2021-005881-17 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease
Keywords: Treprostinil; IPF; ILD
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo inhaled using an ultrasonic nebulizer QID
  Interventions: Drug: Placebo; Device: Treprostinil Ultrasonic Nebulizer
- Inhaled Treprostinil (Experimental): Treprostinil for inhalation solution (0.6 mg/mL) delivered via an ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath. Inhaled QID and titrated up to a target of 12 breaths QID or until the subject reaches their maximum clinically tolerated dose.
  Interventions: Drug: Inhaled Treprostinil; Device: Treprostinil Ultrasonic Nebulizer

INTERVENTIONS:
Drug: Placebo — Placebo administered QID
  Arms: Placebo
Drug: Inhaled Treprostinil — Inhaled treprostinil (6 mcg/breath) administered QID
  Other Names: Tyvaso
  Arms: Inhaled Treprostinil
Device: Treprostinil Ultrasonic Nebulizer — Treprostinil ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath.

SUMMARY:
Study RIN-PF-303 is a multinational study designed to evaluate the superiority of inhaled treprostinil against placebo for the change in absolute forced vital capacity (FVC) from baseline to Week 52.

DETAILED DESCRIPTION:
Study RIN-PF-303 is a multinational, randomized, double-blind, placebo-controlled study to evaluate the superiority of inhaled treprostinil against placebo for the change in absolute FVC in subjects with IPF over a 52-week period. Subjects will be randomly allocated 1:1 to receive inhaled treprostinil or placebo. All subjects will initiate inhaled treprostinil or placebo at a dose of 3 breaths administered 4 times daily (QID) and will titrate to a target dosing regimen of 12 breaths QID. Study drug doses may be titrated up as tolerated, until the target dose or maximum clinically tolerated dose is achieved. Once eligible, 6 Treatment Period visits to the clinic will be required at Weeks 4, 8, 16, 28, 40, and 52.

Efficacy assessments include spirometry (FVC), time to clinical worsening, time to first acute exacerbation of IPF, overall survival, King's Brief Interstitial Lung Disease (K-BILD) questionnaire, plasma N-terminal pro-brain natriuretic peptide (NT-proBNP) concentration, supplemental oxygen use, and lung diffusion capacity (DLCO). Safety assessments include the development of adverse events (AEs)/serious adverse events (SAEs), vital signs, clinical laboratory parameters, and electrocardiogram (ECG) parameters.

Subjects who complete the Week 52 Visit may be offered the opportunity to enter an open-label extension (OLE) study after completing the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject gives voluntary informed consent to participate in the study.
2. Subject is ≥40 years of age, inclusive, at the time of signing informed consent.
3. The subject has a diagnosis of IPF based on the 2018 ATS/ERS/JRS/ALAT Clinical Practice Guideline (Raghu 2018) and confirmed by central review of high-resolution computed tomography (HRCT) (performed within the previous 12 months), and if available, surgical lung biopsy.
4. FVC ≥45% predicted at Screening.
5. Subjects on pirfenidone or nintedanib must be on a stable and optimized dose for ≥30 days prior to Baseline. Concomitant use of both pirfenidone and nintedanib is not permitted.
6. Women of childbearing potential must be non-pregnant (as confirmed by a urine pregnancy test at Screening and Baseline) and non-lactating, and will abstain from intercourse (when it is in line with their preferred and usual lifestyle) or use 2 medically acceptable, highly effective forms of contraception for the duration of the study, and at least 30 days after discontinuing study drug.
7. Males with a partner of childbearing potential must use a condom for the duration of treatment and for at least 48 hours after discontinuing study drug.
8. In the opinion of the Investigator, the subject is able to communicate effectively with study personnel, and is considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.

Exclusion Criteria:

1. Subject is pregnant or lactating.
2. Subject has primary obstructive airway physiology: FEV1/FVC <0.70 at Screening.
3. The subject has shown intolerance or significant lack of efficacy to a prostacyclin or prostacyclin analogue that resulted in discontinuation or inability to effectively titrate that therapy.
4. The subject has received any PAH-approved therapy, including prostacyclin therapy (epoprostenol, treprostinil, iloprost, or beraprost; except for acute vasoreactivity testing), IP receptor agonists (selexipag), endothelin receptor antagonists, phosphodiesterase type 5 inhibitors (PDE5-Is), or soluble guanylate cyclase stimulators within 60 days prior to Baseline. As needed use of a PDE5-I for erectile dysfunction is permitted, provided no doses are taken within 48 hours of any study-related efficacy assessments.
5. Use of any of the following medications: azathioprine (AZA), cyclosporine, mycophenolate mofetil, tacrolimus, oral corticosteroids (OCS) >20 mg/day or the combination of OCS+AZA+N-acetylcysteine within 30 days prior to Baseline; cyclophosphamide within 60 days prior to Baseline; or rituximab within 6 months prior to Baseline.
6. The subject is receiving >10 L/min of oxygen supplementation by any mode of delivery at rest at Baseline.
7. Exacerbation of IPF or active pulmonary or upper respiratory infection within 30 days prior to Baseline. Subjects must have completed any antibiotic or steroid regimens for treatment of the infection or acute exacerbation more than 30 days prior to Baseline to be eligible. If hospitalized for an acute exacerbation of IPF or a pulmonary or upper respiratory infection, subjects must have been discharged more than 90 days prior to Baseline to be eligible.
8. Uncontrolled cardiac disease, defined as myocardial infarction within 6 months prior to Baseline or unstable angina within 30 days prior to Baseline.
9. In the opinion of the Investigator, the subject has any condition that would interfere with the interpretation of study assessments or would impair study participation or cooperation.
10. Use of any other investigational drug/device or participation in any investigational study in which the subject received a medical intervention (ie, procedure, device, medication/supplement) within 30 days prior to Screening. Subjects participating in non-interventional, observational, or registry studies are eligible.
11. Life expectancy <6 months due to IPF or a concomitant illness.
12. Acute pulmonary embolism within 90 days prior to Baseline.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Absolute FVC from Baseline to Week 52 | Baseline to Week 52
  The FVC measurement indicates the amount of air a person can forcefully and quickly exhale after taking a deep breath.

SECONDARY OUTCOMES:
Time to Clinical Worsening | Baseline to Week 52
  Clinical worsening was monitored from randomization until 1 of the following criteria were met: death (all causes), hospitalization due to a respiratory indication, or 10% relative decline in % predicted FVC.
Time to First Acute Exacerbation of IPF | Baseline to Week 52
  An exacerbation of IPF is defined as an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality.
Overall Survival at Week 52 | Baseline to Week 52
  Vital status will be assessed for all subjects at Week 52, including those who discontinue the study prematurely or who withdraw consent.
Change in % Predicted FVC from Baseline to Week 52 | Baseline to Week 52
  The FVC measurement indicates the amount of air a person can forcefully and quickly exhale after taking a deep breath. Percent predicted FVC is calculated based on factors such as ethnicity, sex, age, height, and weight.
Change in K-BILD Questionnaire Score from Baseline to Week 52 | Baseline to Week 52
  The K-BILD is a self-administered, 15-item questionnaire validated for patients with interstitial lung disease (ILD) consisting of 3 domains (breathlessness and activities, psychological, and chest symptoms).
Change in DLCO from Baseline to Week 52 | Baseline to Week 52
  The DLCO measurement measures how well oxygen moves from the lungs to the blood.

CONTACTS AND LOCATIONS:
Locations (108):
- Argentina (9):
  - CINME S.A. - Centro de Investigaciones Metabolicas, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Medico Dra. De Salvo, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Ave Pulmo - Fundación enfisema, Mar del Plata, Buenos Aires
  - Sanatorio Allende S.A., Córdoba, Córdoba Province
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Centro Médico INSARES, Mendoza, Mendoza Province
  - Sanatorio Parque - Consultorios Externos, Rosario, Santa Fe Province
  - Centro Integral de Medicina Respiratoria, San Miguel de Tucumán, Tucumán Province
  - Investigaciones en Patologías Respiratorias, San Miguel de Tucumán, Tucumán Province
- Australia (12):
  - Royal Prince Alfred Hospital, Missenden Road, Camperdown, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Westmead Hospital, Corner of Hawkesbury and Darcy Road, Westmead, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - Lung Research Qld, Chermside, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Respiratory Clinical Trials Pty Ltd, Kent Town, South Australia
  - Alfred Health, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Institute for Respiratory Health - Midland, Nedlands, Western Australia
  - Institute for Respiratory Health - Nedlands, Nedlands, Western Australia
- Belgium (8):
  - Hôpital Erasme, Anderlecht, Brussels Capital
  - CHU UCL Namur asbl - Site Godinne, Yvoir, Namur
  - AZORG vzw, Aalst
  - Ziekenhuis Aan de Stroom, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - CHR de la Citadelle, Liège
  - CHU de Liège, Liège
- Chile (4):
  - Centro de Investigacion del Maule SpA, Talca, Maule Region
  - Oncocentro APYS, Viña del Mar, Región de Valparaíso
  - Instituto Nacional Torax, Santiago, Santiago Metropolitan
  - Fundación Médica San Cristobal, Santiago, Santiago Metropolitan
- Denmark (3):
  - Aarhus University Hospital - Department of Respiratory Diseases and Allergy, Research Unit, Aarhus N
  - Gentofte Hospital - Lungemedicinsk forskning, Hellerup
  - Odense University Hospital - Department of Respiratory Medicine J., Odense C
- France (13):
  - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Hôpital Avicenne, Bobigny, Seine-Saint Denis
  - CHU Amiens Picardie Site Sud - Service de Pneumologie, Amiens
  - Hopital Cote de Nacre, Caen
  - Groupement Hospitalier EST, Service de Pneumologie, Lyon
  - APHM-Hôpital Nord, Marseille
  - Service de Pneumologie, Hôpital Européen Georges Pompídou (HEGP), Paris
  - Hôpital Bichat, Paris
  - CHU Reims - Hôpital Maison Blanche, Reims
  - Hôpital Charles Nicolle-1 Rue de Germont, Rouen
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - Hôpital Larrey, Toulouse
  - CHRU Tours - Hôpital Bretonneau, Tours
- Germany (6):
  - Klinik Löwenstein GmbH, Löwenstein, Baden-Wurttemberg
  - RoMed Klinikum Rosenheim, Rosenheim, Bavaria
  - Universitätsmedezin Essen Ruhrlandklinik Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen, North Rhine-Westphalia
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Fachkrankenhaus Coswig, Coswig
  - LMU Klinikum der Universität, München
- Israel (10):
  - Meir Medical Center, Kfar Saba, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Lady Davis Carmel Medical Center, Haifa, Haifa District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
  - Tel Aviv Sourasky Medical Center - PPDS, Tel Aviv, Southern District
  - Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center - PPDS, Haifa
  - Rabin Medical Center - PPDS, Petah Tikva
- Italy (8):
  - Presidio Ospedaliero GB Morgagni L Pierantoni, Forlì, Emilia-Romagna
  - Ospedale S. Giuseppe Multimedica, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Policlinico "G.Rodolico-San Marco", Catania, Sicily
  - Azienda Ospedaliera Universitaria Senese, Siena, Tuscany
  - Azienda Ospedaliero-Universitaria delle Marche, Ancona
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena
  - Fondazione Policlinico Universitario A Gemelli-Rome, Roma
  - Fondazione PTV Policlinico Tor Vergata, Rome
- Mexico (3):
  - Instituto Nacional De Enfermedades Respiratorias Ismael Cosio Villegas, Mexico City, Mexico City
  - Unidad de Investigación Clínica en Medicina, S.C., Monterrey, Nuevo León
  - Hospital Universitario "Dr. José Eleuterio González", Monterrey, Nuevo León
- Netherlands (3):
  - Zuyderland Medisch Centrum, Heerlen, Limburg
  - Erasmus MC, Rotterdam, South Holland
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
- New Zealand (2):
  - Canterbury Respiratory Research Group, Christchurch, Canterbury
  - Respiratory Medicine, Hamilton, Waikato Region
- Peru (4):
  - Hospital Nacional Adolfo Guevara Velasco, Wanchaq, Departamento de Cusco
  - Clinica Ricardo Palma, Lima, Lima Province
  - Hospital de Chancay y Servicios Basicos deSalud, Huaral, Lima region
  - Hospital Central de la Fuerza Aerea Del Peru, Lima
- South Korea (8):
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - SMG - SNU Boramae Medical Center, Seoul, Seoul Teugbyeolsi
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea - Eunpyeong St. Mary's Hospital, Seoul
  - Samsung Medical Center - PPDS, Seoul
- Spain (11):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Virgen de Las Nieves, Granada, Granada
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- Taiwan (4):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City, Samin District
  - E-DA hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No